CLINICAL TRIAL: NCT01415310
Title: Quality Register for Geriatric Psychiatry in Viken Research Network for Geriatric Psychiatry
Brief Title: Quality Register for Geriatric Psychiatry
Acronym: KVALAP
Status: Recruiting | Type: Observational
Sponsor: Geir Selbaek (Other)
Collaborators: Oslo University Hospital (Other); University Hospital, Akershus (Other); Diakonhjemmet Hospital (Other)
Responsible Party: Sponsor-Investigator, Geir Selbaek, Director of research, Norwegian Centre for Ageing and Health
Organization: Norwegian Centre for Ageing and Health (Other)
Other Study IDs: KVALAP (QualGeP)
Record Dates: First submitted 2011-08-10; First posted 2011-08-11 (Estimated); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Geriatric Disorder; Depression
Keywords: Geriatric Psychiatry; Quality register; Quality improvement; Quality control; Research elderly patients with psychiatric disorders
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Geriatric psychiatry: Elderly patients with psychiatric disorders in geriatric psychiatry units

SUMMARY:
QualGeP (KVALAP) is a quality register in Viken Research network for Geriatric Psychiatry. The objectives of the register are to enhance our knowledge of old persons with severe psychiatric disorders, and to secure an optimal medical evaluation, treatment and care for these patients. The data in the register will be used for quality assurance and for research.

Aims:

* Quality assurance
* Further development of our diagnostic and screening tools
* Contributing to improving the treatment, with and without drugs
* Contributing to improving the dialogue and collaboration between primary healthcare and hospitals

DETAILED DESCRIPTION:
Data collected:

* Demographic data
* Previous and present disorders and use of drugs
* Data from relatives regarding:

  * the patient's cognition
  * psychiatric health
  * behaviour
  * activities of daily living
  * the stress and care burden of relatives
* Tests of cognitive functions
* Methods and duration for treatment
* Transfer to primary healthcare
* Possible readmissions

ELIGIBILITY:
Inclusion Criteria:

* Patients submitted to geriatric psychiatry units and their relatives who sign the consent form

Exclusion Criteria:

* Patients and relatives who refuse to sign the consent form

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients submitted to the geriatric psychiatry units in the Viken Research network for Geriatric Psychiatry
Sampling Method: Non-Probability Sample
Enrollment: 19000 (Estimated)
Dates: Start 2011-04; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Depression and cognition | During admission
  Scores on assessment scales (MADRS, Cornell scale, MMSE)

CONTACTS AND LOCATIONS:
Overall Officials: Knut A. Engedal, professor, Principal Investigator — Norwegian Centre for Ageing and Health
Locations (1):
- Old Age Psychiatry Unit, Diakonhjemmet Hospital, Oslo, Norway